CLINICAL TRIAL: NCT03001050
Title: Rotator Cuff: Does the Vascularity Matter and the Role for PINPOINT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator requested to close, lack of equipment available.
Sponsor: Nirav Amin, MD (Other)
Responsible Party: Sponsor-Investigator, Nirav Amin, MD, M.D. Associate Professor, Loma Linda University
Organization: Loma Linda University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5160379
Record Dates: First submitted 2016-12-05; First posted 2016-12-22 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PINPOINT system (Other): The operative intervention will proceed as current standard protocol dictates for the described procedure. No changes in the operative technique will be undertaken apart from injection of the dye and visualization with the camera. The idea would be to place the Pinpoint probe within the subacromial space, to check the vascular status of the tendon, and then take a bite of the tendon and place the pinpoint back to check if the vascularity has decreased. The Indocyanine Green dye kit will be used along with the PINPOINT system .
  Interventions: Device: PINPOINT System

INTERVENTIONS:
Device: PINPOINT System — To use the camera probe and identify the tendon and footprint vascularity at the time of surgery

SUMMARY:
The overall goal of doing this study is to improve long term patient function and outcomes in the healing rates of Rotator Cuffs. The investigators would also like to see if this method can be more cost effective and time efficient for Rotator Cuff evaluation during arthroscopy.

DETAILED DESCRIPTION:
Background or rationale for this study:

4.5 million Patient's seek medical care for shoulder pain annually in the United States.

250,000 patients receive rotator cuff surgery in the United States annually. Those rotator cuff surgeries produce a societal savings of $3.44 billion per year; averaging $13,771.00 per patient younger than age 61. In which case rotator cuff tears Increases with age.

The Societal and Economic Value of Rotator Cuff Repair (AAOS) 2015 Rotator cuff repairs result in a lifetime societal savings in the U.S. of approximately $3.44 billion annually. Societal savings offset the direct costs of treatment in patients younger than age 61, resulting in an average net savings of $13,771 per patient. This number significantly increased to $77,662.00 for patients younger than 40 years of age.

Common problem, a 55 year-old man injured his left arm. He uses a sling and has difficulties performing simple activities. 1 week later he falls develops immediate pain in his shoulder. On examination he is unable to move his left arm in any upward or sideways direction without supporting it with his other arm. Radiographs he brought show no signs of shoulder osteoarthritis, dislocation, or fracture.

Shoulder pain is the third most common musculoskeletal reason for seeking medical care. Although smaller tears are less likely to propagate, larger tears tend to progress with time and eventually may become irreparable because of significant tendon retraction, muscle atrophy, or both or when the tendons tissue quality does not allow repair.

In 1972-Neer proposed that 95% of rotator cuff injuries were caused by mechanical compression under the coracoacromial arch, others argued cuff tear caused spur formation.

* Type I-flat
* Type II-curved
* Type III-hooked

Multifactorial:

Extrinsic factors;

* Subacromial impingement
* Glenohumeral instability
* Internal impingement
* Trauma (acute/repetitive) Intrinsic Factors;
* Tendon vascular supply
* Collagen fiber abnormalities

A positive painful arc test result and positive external rotation resistance test result were the most accurate finding for detecting Rotator Cuff Disease; whereas the presence of a positive lag tests (external or internal rotation) result was most accurate for diagnosis of a full-thickness rotator cuff tear. Differentiating a full thickness tear from a partial tear, the most sensitive test was the belly-press test (56.8%), and the most specific was the lift-off test (96.95).

Bone microvascularization of the footprint plays a role in rotator Cuff healing. The use of the Pinpoint may play a pivotal role in rotator Cuff healing, en lieu of Plasma Rich platelets with variable results based on concentration levels.

6 level randomized controlled trials showed no clinically significant differences in Constant scores, University of California, Los Angles shoulder rating (UCLA), and American Shoulder and Elbow Surgeons (ASES) scores between double-row and single-row rotator cuff repair. Overall odds ratio (OR) of intact rotator cuff tendon healing was 1.93 in patients treated with double-row versus single-row repair, and the difference was significant.

A statistically significant benefit of double-row repair in the ASES and UCLA scores was observed in the subgroup with tears greater than 3cm. The take home point; Double row may improve structural healing: Clinical Relevance?

9 studies in the meta-analysis, 5 of which were randomized prospective studies (LEVEL1).

Double-row rotator cuff repair techniques have a significantly lower re-tear rate, higher ASES score and greater range of motion of internal rotation compared with single-row repair techniques. Point: Especially in those rotator cuff tears with a size >30mm, the double-row technique is recommended for repair.

This was a Level 4 study out of the Cleveland Clinic which showed the majority of the tears occurred between 6 and 24 weeks. The role of a potential hand held device can assess the tendon quality in the office and change the rehab protocols based on tendon retraction.

Role for study interventions:

* Assessing the bony vascularity at the footprint and the tendon integrity.
* Current standard of care:

Steroid injection as a non-operatively treatment option. Could the steroid injections be affecting the tendon micro vascularization? Could using the Pinpoint assess tendon quality and long term healing a potential.

* Cystic osseous resorption and osteolysis.
* Breakdown products (PLLA) cause synovitis and chondrolysis.
* Breakdown products (PLLA) may interfere with healing-Complications of Bioabsorbable Suture anchors in the shoulder.

Why Medical Row Knots?

* Enhances Biology be sealing footprint from synovial fluid.
* Compared to knotless medical row, better biomechanics incl. load to failure, stiffness, less gap formation.
* A biomechanical comparison of 2 technical of double-row rotator cuff fixation: the importance of medical row knots.

Clinical Implications and Surgeon's Role;

* Choice of a tissue-penetrating instrument; smaller penetrating devices resulting in improves characteristics of stitch holding strength.
* Size of the tissue bite; bigger bite size being stronger.
* Most critical variable under a surgeons control during a rotator cuff repair is the choice of the stitch.

Role for Pinpoint:

In the re-tear and partial-repair groups, postoperative tendon preservation at the middle fact significantly affected the Japanese Orthopaedic Assocation (JOA) and UCLA scores (P=.014, respectively). Considering the patients with tendon healing had better clinical factors, the Pinpoint may help identify the tendon and footprint vascularity at time of surgery.

Goals for the Pinpoint:

To attempt to show that increased vascularity may have an effect of the muscle quality, therefore improving the strength and function long term.

Objective:

* This prospective study aims to obtain the accurate level within a range of a 95% CI imaging Rotator Cuff tendons and the footprint.
* Ensure the Vascularity of the tendon after the footprint and the tendon have been restored to the anatomic footprint. See if the level of the Rotator Cuff bite affects the vascular flow of the tendon.
* Does tying the medical row or excessive tension change the vascularity of the Rotator Cuff.
* We would like to see if by using the Pinpoint system it may be more cost effective then Plasma Rich Platelet.
* Decrease the number of the re-tear rates in Rotator cuff repairs.

Overall goals: Improve long term patient function and outcomes. Increase Rotator Cuff healing rates. Cost effective and time efficient method of Rotator Cuff evaluation during arthroscopy.

Procedures involved (Research Interventions)

Patients undergoing a Rotator Cuff Repair:

* Pre-operatively Questioners to be completed at pre-op American Shoulder and Elbow Surgeons (ASES), University California Los Angeles (UCLA), Disabilities of the arm, shoulder and hand (DASH), Short Form Health Survey-12 (SF-12) & Short Form Health Survey-36 (SF-36)
* Operative Collect OR information
* Post-operative ASES, UCLA, DASH SF-12 & SF-36
* Ultra sounds 3 months, 6 months, 1 year and 24 months

The operative intervention will proceed as current standard protocol dictates for the described procedure. No changes in the operative technique will be undertaken apart from injection of the dye and visualization with the camera. The idea would be to place the Pinpoint probe within the subacrominal space, to check the vascular status of the tendon, and then take a bite of the tendon and place the pinpoint back to check if the vascularity has decreased. The Indocyanin Green dye kit will be used along with the PINPOINT system . Patients with potential allergies or a history of allergies or sensitivity to sodium iodide or iodinated contrast agents should not use this system, and will not be asked to participate. The possible adverse reactions are, anaphylaxis, Hypotension, tachycardia, dyspnea and urticarial. The duration of the procedure will be increased because of the study imaging; this could be 15 to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of requiring Rotator Cuff repair surgical treatment
2. Willingness and ability to comply with the requirements of the protocol including follow-up requirements.
3. Willing and able to sign a study specific informed consent form to participate.
4. Age range of ≥ 30 years old and ≤ 80 years old at time of surgery.
5. Male or female.

Exclusion Criteria:

1. Previous Rotator cuff repair or shoulder surgery.
2. Active systemic infection or infection at the operative site.
3. Co-morbid medical conditions of the upper extremities that may affect the neurological and/or pain assessment.
4. History of an osteoporotic fracture.
5. History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism.
6. Taking medications that may interfere with bony/soft tissue healing including chronic steroid use.
7. Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia.
8. Insulin-dependent type 1 or type 2 diabetes.
9. Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion.
10. Pregnant, or intend to become pregnant, during the course of the study.
11. Severe obesity (Body Mass Index > 40).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
PINPOINT System-ASES | Change from baseline at 24 months
  American Shoulder and Elbow Surgeons questionnaire this will be used for scoring

SECONDARY OUTCOMES:
PINPOINT System-UCLA | Change from baseline at 24 months
  University California Los Angeles, shoulder rating scale
PINPOINT System-DASH | Change from baseline at 24 months
  Disabilities of the arm, shoulder and hand scores
PINPOINT System-SF-36 | Change from baseline at 24 months
  The short form heath survey with 36 questions to measure health status
PINPOINT System-SF-12 | Change from baseline at 24 months
  Short Form Health Survey with 12 questions to measure mental and physical status

CONTACTS AND LOCATIONS:
Overall Officials: Nirav H Amin, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Department of Orthopaedic Surgery, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No